CLINICAL TRIAL: NCT06028490
Title: The Efficacy and Safety of IL4Rα Monoclonal Antibody in Patients With Uncontrolled Seasonal Allergic Rhinitis Under Conventional Treatment: A Randomized, Double-Blind, Placebo-controlled Investigator Initiated Trial.
Brief Title: A Study of IL4Rα Monoclonal Antibody in Patients With Uncontrolled Seasonal Allergic Rhinitis.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zheng Liu ENT (Other)
Responsible Party: Sponsor-Investigator, Zheng Liu ENT, Head of Otolaryngology, Principal Investigator, Clinical Professor, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2081-IIT-SAR
Record Dates: First submitted 2023-08-31; First posted 2023-09-08 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interleukin-4 receptor responders 1 (Experimental): Recombinant fully human anti-IL4Rα monoclonal antibody drug.
  Interventions: Biological: GR1802 injection-1
- Interleukin-4 receptor responders 2 (Experimental): Recombinant fully human anti-IL4Rα monoclonal antibody drug.
  Interventions: Biological: GR1802 injection-2
- Placebo (Placebo Comparator): Recombinant fully human anti-IL4Rα monoclonal antibody drug.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: GR1802 injection-1 — subcutaneous，dose*1
  Other Names: Xeligekimab
  Arms: Interleukin-4 receptor responders 1
Biological: GR1802 injection-2 — subcutaneous，dose*2
  Other Names: Xeligekimab
  Arms: Interleukin-4 receptor responders 2
Biological: Placebo — subcutaneous，dose*2
  Arms: Placebo

SUMMARY:
Allergic rhinitis (AR) is a non-infectious chronic inflammatory disease of the nasal mucosa mainly mediated by immunoglobulin E after exposure to allergens in atopic individuals. The typical symptoms of AR are paroxysmal sneezing, watery rhinorrhea, itching, and nasal congestion, which may be accompanied by ocular symptoms, including eye itching, tearing, redness, and burning sensation, which are more common in patients with hay fever allergies. Bronchial asthma is associated with bronchial asthma in 40% of patients with AR, suggesting a comorbid feature of allergic disease.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects meet the diagnosis of SAR which has been prevalent for at least 2 years, and: standard treatment regimen for SAR was ineffective or subjective symptom control was unsatisfactory in the subject; positive test for at least one allergen associated with the development of SAR; pre-baseline symptom episodes of ≥ 4 days/week and a baseline TNSS of ≥ 6 points.
2. Consent to highly effective contraception

Key Exclusion Criteria:

1. Other nasal comorbidities or co-morbidities/states that may be present at the time of screening；
2. It is expected that subjects' exposure to allergens in their home or work environments may change significantly during the study period.
3. Patients with asthma requiring stable use of inhaled controlled medications;
4. Previous or current malignant tumor within 5 years prior to screening;
5. Presence of other acute or chronic diseases or abnormal laboratory tests at the time of screening that, in the investigator's assessment, may have a more serious impact on the efficacy or safety assessment of the subject;
6. Live/live attenuated vaccine within 3 months prior to baseline;
7. Subjects with very limited outdoor activity during the daytime, as inferred from their regular daily routine;
8. Unwillingness or inability to comply with the permitted and prohibited medication/treatment specifications of the study, inability to meet the pre-randomization drug elution cycle specified in the protocol;
9. Women who are pregnant or breastfeeding;
10. History of alcohol or drug abuse within 3 months prior to screening.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-09-07 (Actual); Primary Completion 2023-11 (Estimated); Study Completion 2023-11 (Estimated)

PRIMARY OUTCOMES:
Average change from baseline in daily retrospective total nasal symptom score (rTNSS) during treatment period. | week 4
  The Total Nasal Symptom Score (TNSS) is the sum of the four symptom scores of runny nose, nasal congestion, nasal itching, and sneezing, with each symptom scoring from 0 to 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hosptial affiliated to Tongji Medical college of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No